CLINICAL TRIAL: NCT04113538
Title: Exploratory and Descriptive Study Evaluating the Efficacy of Aflibercept in Bimonthly Injections Versus the ''Treat and Extend'' Dosing Regimen
Brief Title: Treat and Extend Analysis Trial With Aflibercept in Wet-AMD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Michel Giunta (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor-Investigator, Michel Giunta, P.I., GOGiunta
Organization: GOGiunta (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GOGIUNTA
Record Dates: First submitted 2019-10-01; First posted 2019-10-02 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Wet Age-related Macular Degeneration
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard (Active Comparator): 2 ml (40 mg/ml) of Eylea solution : loading dose of 3 intravitreal injections every 4 weeks for the first 3 months followed by an injection every 8 weeks until the end of the study
  Interventions: Drug: Aflibercept
- Treat and Extend (Experimental): 2 ml (40 mg/ml) of Eylea solution : loading dose of 3 intravitreal injections every 4 weeks for the first 3 months followed and, until the end of the study, retreatment interval based on disease stability
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Aflibercept — Intraocular injection of 2 ml (40mg/ml)
  Other Names: Eylea

SUMMARY:
This study is a randomized, prospective, exploratory, descriptive, open label, parallel group, post-authorization study designed to describe and evaluate two aflibercept treatment regimens aimed at achieving and maintaining a maximum visual function benefit (i.e., BCVA stability). The goal of the study is to compare two strategies for dosing regimen with aflibercept in wet AMD: the standard regimen (one injection every 8 weeks after 3 monthly loading doses in the treatment of wet age-related macular degeneration) versus the treat and extend protocol (details outlined below in the "Study Design" section) aiming at achieving and maintaining maximum visual acuity benefit while minimizing the number of injections. Patients will be randomized at week 8 (Month 2) in a proportion of 1:2 (Standard treatment : treat and extend treatment). We aim to demonstrate that the Treat and Extend regimen is equivalent or better to the standard fixed interval regimen in terms of change in patients' visual acuity after a year of treatment and that patients in the Treat and Extend arm will receive fewer injections and fewer visits, than their counterparts in the standard regimen arm. The results could be used to generate a base for future controlled-randomized clinical trials on the timing of treatment administration for patients with wAMD.

ELIGIBILITY:
Inclusion Criteria:

* Patient who are able to give written informed consent
* Patients 50 years of age or older
* Patients with a diagnosis of treatmenttreatment-naive CNV secondary to AMD in the study eye, for which aflibercept treatment hashas been prescribed by the treating physician. This includes patients with lesion(s) with less than 50% hemorrhage, less that 50% fibrosis, and/or serious pigment epithelial detachment (PED)
* Patients with best corrected visual acuity score in the study eye between 78 and 19 letters inclusively, using ETDRS visual acuity testing charts at a testing distance of 4 meters (approximate Snellen equivalent of 20/32 to 20/400 at screening)
* Females of childbearing potential must, in the opinion of the Investigator, be using a medically effective method of contraception to prevent pregnancy and agree to use an acceptable method of contraception for the duration of their participation in this study. Effective contraception should be used by subjects during the study and for three months after treatment. Effective methods of contraception include, but are not limited to, (i) condoms (male or female) with or without a spermicidal agent; (ii) diaphragm or cervical cap with spermicide; (iii) intra-uterine device; (iv) hormone-based contraception.

Exclusion Criteria:

* Patients with a structural foveal damage - advanced sub retinal fibrosis or significant geographic atrophy involving the foveal center (lack of morphological reserve) in the study eye
* Patients with confounding severe ocular disease in the study eye (such as uncontrolled glaucoma, diabetic retinopathy likely to be visually significant within 2 years, cataract presumably requiring surgery within 2 years) -vitreous or pre-retinal haemorrhage obscuring the central macula, or presence of rhegmatogenous retinal detachment
* Patients with clinical suspicion of polypoidal choroidal vasculopathy
* Patients with active or suspected ocular per ocular infections in either eye
* Patients with active intraocular inflammation in either eye
* Patients with a known sensitivity to Aflibercept or any component of its formulation
* Patients physically unable to tolerate intravenous fluorescein angiography
* Pregnant or breastfeeding female patients
* Any patient with recent history of new onset cardiac disease or thromboembolic event (within 12 months of Baseline visit)
* Patients having received systemic treatment with any other anti-VEGF therapy 60 days prior to enrollment
* Patients having had any prior treatment in the study eye (Avastin, Lucentis, Visudyne, Ozurdex, external radiation therapy, transpupillary thermotherapy, or any intravitreal injection)
* Concurrent participation in a clinical trial or within 30 days prior to enrollment
* Patients with any other condition which, in the opinion of the principal investigator, would require treatment that would significantly impact the treatment assessments during the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity | from baseline to week 52 (Month 12)
  Change in BCVA as measured in with an ETDRS chart
Injections | from baseline to week 52 (Month 12)
  Number of injections

SECONDARY OUTCOMES:
Treatment-free intervals | from baseline to week 52 (Month 12)
  Treatment frequency and duration of treatment-free intervals applied in the treat and extend dosing regimen arm
Gain of letters | from baseline to week 52 (Month 12)
  Proportion of patients with gain of 5 or more, 10 or more, and 15 or more letters
Loss of letters | from baseline to week 52 (Month 12)
  Proportion of patients with loss of 5 or more, 10 or more, and 15 or more letters

CONTACTS AND LOCATIONS:
Locations (1):
- GOGIUNTA, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No